CLINICAL TRIAL: NCT04898608
Title: The Effect of Intradialytic Exercise on Dialysis Patients' Survival: A Randomized Controlled Trial
Brief Title: The Effect of Exercise on Dialysis Patients' Survival
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA20HD-2-01
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2021-05

CONDITIONS: Kidney Disease, Chronic; End Stage Renal Disease; Hemodialysis
Keywords: mortality; exercise during dialysis; physical function; sarcopenia; hematological parameters
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way.
Who Masked: Outcomes Assessor
Masking Description: The lab tech will be blind to whether the sample under evaluation belongs to the intervention group or the control group. A research project collaborator who is not informed about grouping of participants will obtain outcome measurements of the functional test. Outcome adjudicators, and data analysts will be kept blinded to the allocation. Moreover, all investigators, staff, and participants will be kept masked to outcome measurements and trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The patients will participate in intradialytic exercise 3 times a week for 24 weeks.
  Interventions: Other: Intradialytic Exercise
- Control group (No Intervention): The patients will receive regular care and treatment in every dialysis sessions without any intradialytic exercise.

INTERVENTIONS:
Other: Intradialytic Exercise — Participants will do concurrent exercise (a combination of aerobic exercise and resistance training) for 30-60 minutes during the second hour of their routine hemodialysis sessions.
  To determine the intensity of the prescribed exercise, maximum heart rate is used for aerobic workout and 1RM for resistance protocols.
  Exercises will be performed at a moderate exercise intensity (12-14 on the Borg RPE Scale).
  All protocols are tailor-made based on each individual's needs and physical abilities.
  Arms: Exercise group

SUMMARY:
The purpose of this study is to check if patients' exercise during their dialysis sessions can prevent their early deaths.

DETAILED DESCRIPTION:
Dialysis patients suffer from a number of problems, one of which is reduced ability, decreased functional capacity, and consequently reduced physical capability. Forced inactivity due to immobility in dialysis sessions and the need to rest and relieve fatigue for a few hours after each session cause patients to become more inactive day by day, and according to various studies, inactivity in these patients along with reduced physical capabilities increase the risk of cardiovascular disease, which is a risk factor for mortality in these patients.

On the other hand, inactivity is an independent predictor of hospitalization and mortality in these patients.

Studies have shown that exercise can produce many different effects in these patients. However, exercise interventions are often short-term, and even in long-term cases, the aim of studies is only to examine a number of hematological factors or factors such as functional capacity in these patients.

A study is currently being designed to directly evaluate the impact of exercise on patients' survival.

To test this hypothesis, patients do exercise for 6 months during dialysis. And then will be monitored for a year to determine patients' survival.

During 6 months of intervention, hematological parameters, nutrition index and functional capacity of patients are evaluated.

In the analyzes, the survival rate of patients in one year follow-up period is compared between patients who took part in intradialytic sessions (intervention group) and patients who did not do any physical activity during dialysis (control group). In addition, by analyzing the variables measured during the 6 months of the intervention, the effect of exercise on parameters relating to survival is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis history ≥ 1 year
* Without myocardial infarction within past 3 months
* Regular dialysis 3 times a week
* Ability to consent
* Doctor's consent

Exclusion Criteria:

* Unstable cardiac status (angina, decompensated congestive heart failure, severe arteriovenous stenosis, uncontrolled arrhythmias, etc.)
* Active infection or acute medical illness
* Hemodynamic instability
* Labile glycemic control
* Unable to exercise (lower extremity amputation with no prosthesis)
* having severe musculoskeletal pain at rest or with minimal activity
* Unable to sit, stand or walk unassisted (walking device such as cane or walker allowed)
* Having shortness of breath at rest or with activities of daily living (NYHA Class IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
1-year Survival of dialysis patients | Follow-up phase (1- year)
  Mortality data is gathered using form "CMS-2746" which is specifically for dialysis patients.

SECONDARY OUTCOMES:
Rate of changes of Albumin for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Hemoglobin for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Hematocrit for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Red Blood Cells for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Calcium for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Phosphorus for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Parathyroid Hormone for 6 months | Pre_test and every 3 months for 6 months
Changes of GNRI for 6 months | Pre_test and every 3 months for 6 months
  The Geriatric Nutritional Risk Index (GNRI) is a screening method that was primarily developed to identify older patients with malnutrition. It consists of serum albumin levels as well as body weight measurements. GNRI is associated with an increasing risk of long-term all-cause mortality in prevalent hemodialysis patients, even after adjusting for age and comorbidity
Changes of the meters walked during the 6MWT for 6 months | Pre_test and every 3 months for 6 months
  Six-minute walk test (6MWT) is a walking endurance assessment measured in meters of total distance completed over 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Principal Investigator — Pardis Specialized Wellness Institute
Locations (2):
- Iran (2):
  - Abolfazl medical center, Isfahan
  - Pardis specialized wellness institute, Isfahan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification are to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: The IPD will be available only for our colleagues in GREX as long as they have acceptable reasons for requiring the data.

REFERENCES:
- [Background] Xiong J, Wang M, Zhang Y, Nie L, He T, Wang Y, Huang Y, Feng B, Zhang J, Zhao J. Association of Geriatric Nutritional Risk Index with Mortality in Hemodialysis Patients: A Meta-Analysis of Cohort Studies. Kidney Blood Press Res. 2018;43(6):1878-1889. doi: 10.1159/000495999. Epub 2018 Dec 14. PMID 30566933
- [Background] Tabibi MA, Ahmadi E, Nasrin S. POS-621 The effect of concurent exercise during dialysis on hemoglobin,red blood cells and hematocrit in hemodialysis patients. Kidney International Reports. 2021; 6(4): 270-271. doi: 10.1016/j.ekir.2021.03.650
- [Background] Shimoda T, Matsuzawa R, Yoneki K, Harada M, Watanabe T, Matsumoto M, Yoshida A, Takeuchi Y, Matsunaga A. Changes in physical activity and risk of all-cause mortality in patients on maintence hemodialysis: a retrospective cohort study. BMC Nephrol. 2017 May 8;18(1):154. doi: 10.1186/s12882-017-0569-7. PMID 28482880
- [Background] Bakaloudi DR, Siargkas A, Poulia KA, Dounousi E, Chourdakis M. The Effect of Exercise on Nutritional Status and Body Composition in Hemodialysis: A Systematic Review. Nutrients. 2020 Oct 8;12(10):3071. doi: 10.3390/nu12103071. PMID 33050111
- [Background] Parker K. Intradialytic Exercise is Medicine for Hemodialysis Patients. Curr Sports Med Rep. 2016 Jul-Aug;15(4):269-75. doi: 10.1249/JSR.0000000000000280. PMID 27399824
- [Background] K/DOQI Workgroup. K/DOQI clinical practice guidelines for cardiovascular disease in dialysis patients. Am J Kidney Dis. 2005 Apr;45(4 Suppl 3):S1-153. No abstract available. PMID 15806502
- [Background] Milam RH. Exercise Guidelines for Chronic Kidney Disease Patients. J Ren Nutr. 2016 Jul;26(4):e23-5. doi: 10.1053/j.jrn.2016.03.001. No abstract available. PMID 27318109
- [Background] Scapini KB, Bohlke M, Moraes OA, Rodrigues CG, Inacio JF, Sbruzzi G, Leguisamo CP, Sanches IC, Tourinho Filho H, Irigoyen MC. Combined training is the most effective training modality to improve aerobic capacity and blood pressure control in people requiring haemodialysis for end-stage renal disease: systematic review and network meta-analysis. J Physiother. 2019 Jan;65(1):4-15. doi: 10.1016/j.jphys.2018.11.008. Epub 2018 Dec 21. PMID 30581137
- [Background] Huang M, Lv A, Wang J, Xu N, Ma G, Zhai Z, Zhang B, Gao J, Ni C. Exercise Training and Outcomes in Hemodialysis Patients: Systematic Review and Meta-Analysis. Am J Nephrol. 2019;50(4):240-254. doi: 10.1159/000502447. Epub 2019 Aug 27. PMID 31454822
- [Background] Pu J, Jiang Z, Wu W, Li L, Zhang L, Li Y, Liu Q, Ou S. Efficacy and safety of intradialytic exercise in haemodialysis patients: a systematic review and meta-analysis. BMJ Open. 2019 Jan 21;9(1):e020633. doi: 10.1136/bmjopen-2017-020633. PMID 30670499
- [Background] Zhang F, Zhou W, Sun Q, Zhai Y, Zhang Y, Su H, Wang Z. Effects of intradialytic resistance exercises on physical performance, nutrient intake and quality of life among haemodialysis people: A systematic review and meta-analysis. Nurs Open. 2021 Mar;8(2):529-538. doi: 10.1002/nop2.274. Epub 2019 Sep 30. PMID 33570280
- [Background] Noordzij M, Korevaar JC, Boeschoten EW, Dekker FW, Bos WJ, Krediet RT; Netherlands Cooperative Study on the Adequacy of Dialysis (NECOSAD) Study Group. The Kidney Disease Outcomes Quality Initiative (K/DOQI) Guideline for Bone Metabolism and Disease in CKD: association with mortality in dialysis patients. Am J Kidney Dis. 2005 Nov;46(5):925-32. doi: 10.1053/j.ajkd.2005.08.013. PMID 16253734
- [Background] Stevens LA, Djurdjev O, Cardew S, Cameron EC, Levin A. Calcium, phosphate, and parathyroid hormone levels in combination and as a function of dialysis duration predict mortality: evidence for the complexity of the association between mineral metabolism and outcomes. J Am Soc Nephrol. 2004 Mar;15(3):770-9. doi: 10.1097/01.asn.0000113243.24155.2f. PMID 14978180
- [Background] Pifer TB, McCullough KP, Port FK, Goodkin DA, Maroni BJ, Held PJ, Young EW. Mortality risk in hemodialysis patients and changes in nutritional indicators: DOPPS. Kidney Int. 2002 Dec;62(6):2238-45. doi: 10.1046/j.1523-1755.2002.00658.x. PMID 12427151
- [Background] Avram MM, Blaustein D, Fein PA, Goel N, Chattopadhyay J, Mittman N. Hemoglobin predicts long-term survival in dialysis patients: a 15-year single-center longitudinal study and a correlation trend between prealbumin and hemoglobin. Kidney Int Suppl. 2003 Nov;(87):S6-11. doi: 10.1046/j.1523-1755.64.s87.3.x. PMID 14531767
- [Background] Foley RN, Parfrey PS, Morgan J, Barre PE, Campbell P, Cartier P, Coyle D, Fine A, Handa P, Kingma I, Lau CY, Levin A, Mendelssohn D, Muirhead N, Murphy B, Plante RK, Posen G, Wells GA. Effect of hemoglobin levels in hemodialysis patients with asymptomatic cardiomyopathy. Kidney Int. 2000 Sep;58(3):1325-35. doi: 10.1046/j.1523-1755.2000.00289.x. PMID 10972697
- [Background] Bohm CJ, Ho J, Duhamel TA. Regular physical activity and exercise therapy in end-stage renal disease: how should we move forward? J Nephrol. 2010 May-Jun;23(3):235-43. PMID 20383863
- [Background] Aucella F, Gesuete A, Battaglia Y. A "nephrological" approach to physical activity. Kidney Blood Press Res. 2014;39(2-3):189-96. doi: 10.1159/000355796. Epub 2014 Jul 29. PMID 25118037
- [Background] Wilund K, Thompson S, Bennett PN. A Global Approach to Increasing Physical Activity and Exercise in Kidney Care: The International Society of Renal Nutrition and Metabolism Global Renal Exercise Group. J Ren Nutr. 2019 Nov;29(6):467-470. doi: 10.1053/j.jrn.2019.08.004. Epub 2019 Oct 4. No abstract available. PMID 31591041
- [Background] Kohl Lde M, Signori LU, Ribeiro RA, Silva AM, Moreira PR, Dipp T, Sbruzzi G, Lukrafka JL, Plentz RD. Prognostic value of the six-minute walk test in end-stage renal disease life expectancy: a prospective cohort study. Clinics (Sao Paulo). 2012;67(6):581-6. doi: 10.6061/clinics/2012(06)06. PMID 22760895
- [Background] Evangelidis N, Tong A, Manns B, Hemmelgarn B, Wheeler DC, Tugwell P, Crowe S, Harris T, Van Biesen W, Winkelmayer WC, Sautenet B, O'Donoghue D, Tam-Tham H, Youssouf S, Mandayam S, Ju A, Hawley C, Pollock C, Harris DC, Johnson DW, Rifkin DE, Tentori F, Agar J, Polkinghorne KR, Gallagher M, Kerr PG, McDonald SP, Howard K, Howell M, Craig JC; Standardized Outcomes in Nephrology-Hemodialysis (SONG-HD) Initiative. Developing a Set of Core Outcomes for Trials in Hemodialysis: An International Delphi Survey. Am J Kidney Dis. 2017 Oct;70(4):464-475. doi: 10.1053/j.ajkd.2016.11.029. Epub 2017 Feb 24. PMID 28238554
- [Background] Chantrel F, de Cornelissen F, Deloumeaux J, Lange C, Lassalle M; registre REIN. [Survival and mortality in ESRD patients]. Nephrol Ther. 2013 Sep;9 Suppl 1:S127-37. doi: 10.1016/S1769-7255(13)70042-7. French. PMID 24119578
- [Derived] Tabibi MA, Cheema B, Salimian N, Correa HL, Ahmadi S. The effect of intradialytic exercise on dialysis patient survival: a randomized controlled trial. BMC Nephrol. 2023 Apr 17;24(1):100. doi: 10.1186/s12882-023-03158-6. PMID 37069527